CLINICAL TRIAL: NCT00002455
Title: Immunotherapy of Colon Cancer With Autologous Perchloric Soluble Tumors Extracts
Brief Title: Immunotherapy After Surgery in Treating Patients With Breast Cancer, Colon Cancer, or Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Oncologico de Excelencia (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: ARG-CO/BR-1; CDR0000072435 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 1998-11

CONDITIONS: Breast Cancer; Colorectal Cancer; Melanoma (Skin)
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; recurrent breast cancer; recurrent colon cancer; stage I melanoma; stage II melanoma; stage III melanoma; recurrent melanoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Melanoma; Colonic Neoplasms | interventions — Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: Corynebacterium granulosum P40
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Immunotherapy uses different ways to stimulate the immune system and stop cancer cells from growing. Immunotherapy biological extracts may be useful as adjuvant therapy in treating patients who have had surgery for breast cancer, colon cancer, or melanoma.

PURPOSE: Phase III trial to study the effectiveness of Corynebacterium granulosum extract as maintenance immunotherapy following surgery in treating patients with breast cancer, colon cancer, or melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the survival of patients with colon cancer, breast cancer, or melanoma with minimal residual disease after surgical resection treated with maintenance immunotherapy using Corynebacterium granulosum P40.
* Determine leucocyte adherence inhibition, an indication of metastases, over time in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified by center and are matched with case-controls by disease type and stage.

Beginning 2 weeks after surgical resection, patients receive Corynebacterium granulosum P40 subcutaneously weekly for 6 weeks, followed by rest for 3 months. Treatment continues for life.

Patients are followed for survival.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colon cancer, breast cancer, or melanoma with minimal residual disease (at least 90% of tumor mass resected) after surgical resection
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 20 to 80

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1971-04

PRIMARY OUTCOMES:
Recurrence
Response to study parameters
Survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Omar De Carli, MD, Study Chair — Centro Oncologico de Excelencia
Locations (1):
- Centro Oncologico de Excelencia, Manuel B. Gonnet, Buenos Aires, Argentina

REFERENCES:
- [Background] De Carli HO: Immunostimulation and follow-up in long term subclinical cancer. Buenos Aires. Argentina: Centro Oncologico de Excelencia.